CLINICAL TRIAL: NCT02643602
Title: Does Bicarbonate in Addition to Theophylline Reduce Contrast Induced Nephropathy Compared to Sodium Chloride?
Brief Title: Does Bicarbonate in Addition to Theophylline Reduce CIN?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NaBicTheo
Record Dates: First submitted 2015-12-23; First posted 2015-12-31 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Radiographic Contrast Agent Nephropathy
MeSH Terms: interventions — Bicarbonates; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bicarbonate and theophylline (Experimental): Hydration with bicarbonate in addition to theophylline
  Interventions: Other: Hydration with bicarbonate in addition to theophylline
- Sodium and theophylline (Active Comparator): Hydration with sodium chloride in addition to theophylline
  Interventions: Other: Hydration with sodium chloride in addition to theophylline

INTERVENTIONS:
Other: Hydration with bicarbonate in addition to theophylline — 0.154-molar sodium bicarbonate; 3 ml per kg bodyweight (maximum 330 ml) one hour before contrast exposure; additionally 200 mg theophylline as a short infusion; after contrast application hydration with another 1 ml per kg bodyweight per hour (maximum 110 ml per hour) for 6 hours
  Arms: Bicarbonate and theophylline
Other: Hydration with sodium chloride in addition to theophylline — 0.9% sodium chloride; 3 ml per kg bodyweight (maximum 330 ml) one hour before contrast exposure; additionally 200 mg theophylline as a short infusion; after contrast application hydration with another 1 ml per kg bodyweight per hour (maximum 110 ml per hour) for 6 hours
  Arms: Sodium and theophylline

SUMMARY:
Contrast-induced nephropathy (CIN) is the third most frequent cause of hospital-acquired acute renal failure. Different regimes in the prophylaxis of CIN have been investigated in the last years. Recent Meta-analysis show a reduced incidence of CIN when theophylline is administered to the patients especially in patients with already existing renal impairment. Furthermore hydration with bicarbonate seems to to be superior to hydration with sodium chloride alone. The combination of the two prophylaxis has not been investigated yet.

Aim of this prospective randomized trial is to investigate the effect of hydration with sodium bicarbonate compared to saline in addition to theophylline prophylaxis which all patients receive.

ELIGIBILITY:
Inclusion Criteria:

Increased risk for contrast induced nephropathy defined as:

* Serum creatinine level ≥ 1.1 mg/dl OR
* Serum creatinine level ≥ 0.8 mg/dl plus an additional risk factor like diabetes mellitus, renal failure in past medical history or nephrotoxic medication (aminoglycoside, vancomycin, amphotericin B, diuretic)

Exclusion Criteria:

* pre-existing renal replacement therapy
* unstable serum creatinine levels (difference of more than ±0.4 mg/dl within 3 days before contrast application)
* contraindications for theophylline or sodium bicarbonate (allergies, tachycardia, alkalosis, hypokalemia)
* additional interventions that might influence renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2005-12; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Contrast induced nephropathy | 48 hours
  Raise in serum creatinine of ≥25% or ≥0.5 mg/dl

SECONDARY OUTCOMES:
Change of serum creatinine levels over time | 48 hours
Change of creatinine clearance over time | 48 hours
Change in blood pH | 48 hours
Change in blood bicarbonate-concentration | 48 hours
Change in blood sodium-concentration | 48 hours
Change in urine pH | 48 hours
Change in urine bicarbonate-concentration | 48 hours
Change in urine pH sodium-concentration | 48 hours
Incidence of patients with need for dialysis | 30 days
  The patients medical record was reviewed to determine whether dialysis was performed within 30 days after contrast media application.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Huber, M.D., Principal Investigator — 2. Medizinische Klinik, Klinikum rechts der Isar der Technischen Universität München